CLINICAL TRIAL: NCT01835106
Title: A Prospective, Randomized, Double-blind, Placebo-controlled, Crossover Trial of Epidural Analgesia Versus a Surgically-placed Fascia Iliaca Compartment Catheter for Postoperative Pain After Periacetabular Osteotomy
Brief Title: Efficacy of an Epidural Versus a Fascia Iliaca Compartment Catheter After Hip Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was proposed but never started due to other commitments
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Luke Y. Wang, Instructor in Anesthesia, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3650
Record Dates: First submitted 2013-04-16; First posted 2013-04-18 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Postoperative Pain
Keywords: Postoperative Care
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Epidural (Active Comparator): Epidural catheter is used postoperatively
  Interventions: Procedure: Epidural catheter is used postoperatively
- Fascia Iliaca Compartment (Experimental): Fascia iliaca compartment catheter is used postoperatively
  Interventions: Procedure: Fascia iliaca compartment catheter is used postoperatively

INTERVENTIONS:
Procedure: Epidural catheter is used postoperatively
  Arms: Epidural
Procedure: Fascia iliaca compartment catheter is used postoperatively
  Arms: Fascia Iliaca Compartment

SUMMARY:
The investigators are investigating two ways of treating pain after hip surgery. One way is though a thin tube (called a catheter), and it is placed into the back so that pain-numbing drugs can reach the nerves near the backbone. This is called an "epidural" catheter. Another way is to place the catheter close to the hip, where the surgery is done, so that the pain-numbing drugs can reach some of the nerves more locally. This is called a "fascia iliaca compartment" catheter.

The investigators do not know which way is best to treat pain, or has fewer side effects, or allows a patient to leave hospital faster. Usually, patients would receive only one type of catheter for pain relief. To do this comparison, the investigators would place both catheter types, so that patients help us tell which one works better.

ELIGIBILITY:
Inclusion Criteria:

* Weight >40 kg
* Radiographic evidence of hip dysplasia amenable to unilateral surgical treatment by periacetabular osteotomy
* Western Ontario and McMaster Universities Arthritis Index (WOMAC) pain subscale >4/20
* Age between 15 and 35 years
* Good or excellent preoperative joint congruency

Exclusion Criteria:

* Hematologic or neurologic contraindications to epidural catheter placement
* Significant renal, hepatic, or cardiac disease
* Peptic ulcer disease
* Bleeding disorders
* Severe asthma
* Hypersensitivity to non-steroidal antiinflammatory drugs
* Developmental delay
* History of substance abuse
* Chronic opioid use
* Chronic pain in non-hip locations

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Number of days until all pre-defined readiness-to-discharge criteria for hip surgery are met | 1-5 days
  1. Numerical pain rating score <4 at rest, and <6 with movement,
  2. Independence from intravenous opioids for 12 hours, and
  3. Ambulation at least 30 m, without a time limit

CONTACTS AND LOCATIONS:
Overall Officials: Luke Y Wang, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States